CLINICAL TRIAL: NCT06944808
Title: Impact of Blood Flow Restriction and Electrical Stimulation on Postoperative Muscle Atrophy and Pain After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Dr. med., B.Sc., University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023_B
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis Knees
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham-BFR + Electrical Stimulation (Active Comparator): Patients received a daily postoperative passive therapy with a sham-BFR intervention (20mmHg) and electrical stimulation of the M. vastus laterals and mediales.
  Interventions: Other: Sham-BFR + EMS
- BFR + Electrical Stimulation (Experimental): Patients received a daily postoperative passive therapy with a BFR intervention (80% of the individual LOP) and electrical stimulation of the M. vastus laterals and mediales.
  Interventions: Other: BFR + EMS

INTERVENTIONS:
Other: Sham-BFR + EMS — Daily passive sham-BFR with a fixed pressure of 20mmHg in combination with electrical stimulation of the m. vastus lateralis and mediales
  Arms: Sham-BFR + Electrical Stimulation
Other: BFR + EMS — Daily passive BFR with an individual pressure of 80% of the limb occlusion pressure in combination with electrical stimulation of the m. vastus lateralis and mediales
  Arms: BFR + Electrical Stimulation

SUMMARY:
This study investigate the impact of Blood Flow Restriction Training and Electrostimulation Training on postoperative muscle atrophy and pain after elective total knee arthroplasty.

DETAILED DESCRIPTION:
The present study invesigate the impact of passive blood flow restriction training and/or electrical stimulation training on postoperative muscle atrophy and pain after elective total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Indication for elective total knee arthroplasty
* Understanding of the study and ability for informed consent

Exclusion Criteria:

* Open wounds of the lower extremities
* Stents or bypasses on the location of pressure application
* Sickle Cell Anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | Pre- to 6 week Post-OP
  Visual Analog Scale (0-100mm)
Muscle Mass | Pre- to 6 week Post-OP
  Sonographic measure of the diameter of the M. vastus mediales and lateralis

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No